CLINICAL TRIAL: NCT06186102
Title: Polyamine Treatment in Elderly Patients With Coronary Artery Disease - a Randomized Controlled Trial
Brief Title: Polyamine Treatment in Elderly Patients With Coronary Artery Disease
Acronym: PolyCAD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Sygesikringen Danmark (Unknown); Steno Diabetes Center Aarhus (SDCA), Aarhus University Hospital (Unknown); Danish Diabetes Academy (Other); Danish Cardiovascular Academy (DCA) (Unknown); Eva and Henry Frænkels Mindefond (Unknown); DoNotAge.org (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-2023-71-23
Record Dates: First submitted 2023-12-07; First posted 2023-12-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Heart Disease; Myocardial Infarction; Cardiovascular Diseases; Hypertensive Heart Disease; Hypertension; Diastolic Dysfunction; Obesity; Metabolic Syndrome; Diabetes Mellitus, Type 2; Dietary Habits; Inflammation; Quality of Life; Cognition Disorder; Cognitive Impairment
Keywords: Spermidine; Dietary supplement; Polyamine; Prevention; Treatment; Lifestyle; Coronary artery disease; Ischemic heart disease; Cardiovascular disease; Heart disease; Hypertension; Obesity; Diabetes Mellitus, Type 2; Insulin resistance; Inflammation; Quality of life; Cognitive function; Memory; Autophagy
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction; Cardiovascular Diseases; Hypertension; Obesity; Metabolic Syndrome; Diabetes Mellitus, Type 2; Feeding Behavior; Inflammation; Cognition Disorders; Cognitive Dysfunction; Coronary Artery Disease; Heart Diseases; Insulin Resistance | interventions — Spermidine; Polyamines

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, two-armed, parallel-group, single centre, clinical study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spermidine (Active Comparator): Spermidine will be given orally as capsules of cellulose with spermidine (24 mg/day) and rice flour.
  Interventions: Dietary Supplement: Spermidine
- Placebo (Placebo Comparator): Placebo will be given orally as capsules of cellulose and rice flour (same size and visual appearance as spermidine capsules)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Spermidine — Spermidine capsule of 8 mg x 3 capsules daily.
  Other Names: Polyamine
  Arms: Spermidine
Other: Placebo — Placebo capsule. 3 capsules daily.
  Arms: Placebo

SUMMARY:
The present study is testing spermidine treatment in elderly patients with coronary artery disease. The study is a randomized, double-blind, placebo-controlled, two-armed, parallel-group, single centre, clinical study.

DETAILED DESCRIPTION:
Life expectancy has increased tremendously over the past century and as populations age, chronic diseases such as cardiovascular disease and diabetes have become more prevalent. Healthy aging is therefore of paramount importance to further promote longevity and quality of life.

In humans, a high concentration of whole-blood spermidine is associated with longevity, and individuals with a high dietary spermidine intake have improved cardiovascular health and less obesity. Spermidine is essentially a polyamine found in all plant-derived foods, particularly in whole grains, soybeans, nuts, and fruit. Its favorable effects may act via several mechanisms. In an experimental model of hypertensive heart disease, spermidine reduced cardiac hypertrophy and improved diastolic and mitochondrial function. Spermidine also induces cytoprotective autophagy in skeletal muscle and alters body fat accumulation by metabolically modulating glucose and lipid metabolism.

The clinical data on spermidine dietary supplementation are scarce. In elderly subjects with cognitive problems, spermidine supplement was well tolerated and had potential blood-pressure-lowering effects. The reported beneficial effects of spermidine raise the question whether elderly patients with cardiovascular disease can benefit from a dietary supplement of this polyamine.

The central hypothesis of the current proposal is that a twelve-month spermidine treatment regimen in elderly patients with cardiovascular disease will yield positive effects on heart and skeletal muscle function, whole body composition and inflammation. The secondary hypotheses are that spermidine reduces blood pressure and has a beneficial impact on cognitive function, daily activity level, quality of life, biomarker risk profile, skeletal muscle cellular metabolism and lastly but not least gut microbiota.

The study design is a randomized, double-blind, placebo-controlled trial to investigate the effects of a 24 mg daily oral spermidine dietary supplement vs. matching placebo in elderly patients with cardiovascular disease. A total of 200 patients will be included and randomized 1:1 to either spermidine 24 mg x 1 daily or matching placebo for one year.

At baseline and after one year of intervention the patients will undergo study procedures. Changes from baseline to follow-up will be compared between the active and placebo treated patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Chronic ischemic heart disease (previous revascularization or myocardial infarction)
* Left ventricular ejection fraction of > 40%

And at least two of the following risk factors:

* Type 2 diabetes,
* Obesity (BMI ≥ 30 kg/m2),
* Hypertension,
* Previous LVEF < 40%,
* Left atrial volume index ≥ 30 mL/m2
* Left ventricular wall thickness ≥ 1.1 cm.

Exclusion Criteria:

* Unstable coronary syndrome
* Significant and severe cardiac valve disease
* Severe peripheral artery disease
* Permanent atrial fibrillation
* Pacemaker treatment
* Chronic kidney disease with eGFR <45 ml/min/1,73m2
* Severe comorbidity as judged by the investigator (such as severe pulmonary, neurological, or musculoskeletal disease)
* Inability to give informed consent.

Exclusion criteria for MRI:

* Some metallic implants
* Claustrophobia

Exclusion criteria for muscle biopsy:

* Treatment with either two antiplatelet drugs (aspirin and ADP-receptor antagonists)
* Anticoagulants (warfarin, NOACs)

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass | From randomization (month 0) to 12 months
  Measured with Cardiac Magnetic Resonance Imaging (CMR).
Change in appendicular lean mass and ALM index | From randomization (month 0) to 12 months
  Appendicular lean mass and ALM index (Appendicular lean mass/height^2). Measured by a whole-body dual-energy X ray absorptiometry (DXA) scan.
Change in High-sensitivity C-reactive Protein (hs-CRP) | From randomization (month 0) to 12 months
  Measured from blood samples.
Change in Physical performance, peak oxygen consumption (VO2max) | From randomization (month 0) to 12 months
  Measured by cardiopulmonary exercise capacity (CPET) will be performed using a cycle ergometer test. Peak oxygen uptake measured in ml O2/kg/min.

SECONDARY OUTCOMES:
Muscle strength, Handgrip strength | From randomization (month 0) to 12 months
  Hand-held dynamometer for measuring handgrip strength in kilograms.
Muscle strength, Knee-extension/flexion strength | From randomization (month 0) to 12 months
  Change in knee extension and flexion isokinetic strength (assessed by peak torque, Nm) and isometric strength (assessed by peak torque, Nm).
Physical performance, 6 minute walk test (6MWT) | From randomization (month 0) to 12 months
  Change in walking distance in meters.
Physical performance, 30 seconds sit to stand test | From randomization (month 0) to 12 months
  Change in counts of sit to stand.
The Short Physical Performance Battery | From randomization (month 0) to 12 months
  Changes in points.
Skeletal muscle mass | From randomization (month 0) to 12 months
  Thigh muscle mass by Magnetic Resonance Imaging (MRI) using Dixon method.
Skeletal muscle cross sectional area (CSA) of fibers | From randomization (month 0) to 12 months
  CSA of fibers by cryosection of skeletal muscle biopsy obtained from vastus lateralis muscle.
Skeletal muscle tissue fiber composition | From randomization (month 0) to 12 months
  Change in ratio between muscle fiber types (type I, IIa and IIb) assessed by immunohistochemistry.
Skeletal muscle tissue cellular composition | From randomization (month 0) to 12 months
  Change in muscle tissue cellular composition assessed by cell sorting
Skeletal muscle mitochondrial function | From randomization (month 0) to 12 months
  Change in muscle mitochondrial function assessed by high-resolution respirometry
Total lean body mass | From randomization (month 0) to 12 months
  Change in lean body mass (in grams) and total lean mass/height^2.
Total body fat percentage | From randomization (month 0) to 12 months
  Changes in body fat percentage.
Estimated visceral adipose tissue | From randomization (month 0) to 12 months
  Change in VAT index (kilogram-per-meters-squared index) and in mass (in grams).
Intramuscular and intermuscular fat content | From randomization (month 0) to 12 months
  Calculating thigh adipose tissue mass located between and within muscle fibers by MRI Dixon method.
Free fatty acids | From randomization (month 0) to 12 months
  Measured from blood samples.
Insulin resistance | From randomization (month 0) to 12 months
  Changes in insulin resistance assessed by Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Markers of autophagy | From randomization (month 0) to 12 months
  Proteomics of skeletal muscle tissue and peripheral blood mononuclear cells (PBMCs).
Polyamine content in muscle biopsy | From randomization (month 0) to 12 months
  Measured with liquid chromatography mass spectrometry (LC-MS).
Polyamine content in blood | From randomization (month 0) to 12 months
  Plasma samples obtained from blood. Measured with liquid chromatography mass spectrometry (LC-MS).
Change in 24-hour ambulatory blood pressure measurements (24h ABPM) | From randomization (month 0) to 12 months
  Measured with the Spacelabs Healthcare 90217A device in an out-of-hospital setting.
Change in central blood pressure | From randomization (month 0) to 12 months
  Measured noninvasive with pulse wave analysis (PWA) using a SphygmoCor system.
Change in daily physical activity | From randomization (month 0) to 12 months
  Assessed by 14-day activity monitoring with an accelerometer (AX3, Axivity).
Change in cardiac extracellular volume fraction | From randomization (month 0) to 12 months
  Assessed using Cardiac Magnetic Resonance Imaging (CMR) with intravenous gadolinium-based agent.
Change in myocardial strain | From randomization (month 0) to 12 months
  Assessed using Cardiac Magnetic Resonance Imaging (CMR) with intravenous gadolinium-based agent.
Change in Carotid-femoral pulse wave velocity | From randomization (month 0) to 12 months
  Measured non-invasively through applanation tonometry using a SphygmoCor system. The unit of measure is m/s.
Change in Aortic pulse wave velocity | From randomization (month 0) to 12 months
  Magnetic resonance imaging (MRI) assessment. The unit of measure is m/s.
Change in general cognitive function and memory performance | From randomization (month 0) to 12 months
  Evaluated using the Montreal Cognitive Assessment (MoCA). It will be administered in a clinical setting using a tablet. MoCA score ranges from 0-30 and a score of 26 or higher is considered normal.
Change in specific domains of cognitive function | From randomization (month 0) to 12 months
  Evaluated using Cambridge Cognition (CANTAB) digital assessment software in a clinical setting using a tablet. The cognitive tests are MOT, RTI, SWM, DMS and PAL. These tests will objectively measure psychomotor speed, executive function and memory.
HeartQol | From randomization (month 0) to 12 months
  HeartQol measures health-related quality of life (HRQL) and is a disease-specific health status instrument for ischemic heart disease. It consists of 14 items and provides two subscales; a 10-item physical subscale and a 4-item emotional subscale, which are scored on a four-point Likert scale (0 to 3). Higher scores indicate a better HRQL. Measured as global, physical and emotional score.
Cytokines | From randomization (month 0) to 12 months
  Changes in cytokines are evaluated through the utilization of multiplex cytokine assays. Measured from plasma blood samples.
White blood cells | From randomization (month 0) to 12 months
  Changes in white blood cell differential count.
Immune cells | From randomization (month 0) to 12 months
  Changes in specific immune cell populations are measured using peripheral blood mononuclear cells (PBMCs) isolated from blood samples.
Vascular inflammatory markers | From randomization (month 0) to 12 months
  Measured from plasma blood samples with a multiplex assay.
Time to first occurrence of Composite cardiovascular endpoint: Cardiovascular death, heart failure hospitalizations, non-fatal myocardial infarction, non-fatal stroke, and coronary revascularization | From randomization (month 0) to 12 months
  Measured in months.
Days alive and out of hospital | From randomization (month 0) to 12 months
  Measured in months.

OTHER OUTCOMES:
Changes in gut microbiota | From randomization (month 0) to 12 months
  16S RNA analysis will be used for characterization of the bacterial composition.
  Full sequencing will be used for characterisation of the collective composition of bacteria, viruses, bacteriophages, fungi, and parasites.
Changes in fecal metabolites | From randomization (month 0) to 12 months
  Mass spectrometric metabolome analyses will be used for assessing fecal metabolites before and after intervention.
Skeletal muscle quality assesment | From randomization (month 0) to 12 months
  An explorative analysis of skeletal muscle quality including MRI with Dixon method, fiber CSA and type composition, tissue vascularity, morphology and architecture of skeletal muscle biopsy taken from vastus lateralis.
Explorative analysis of adipose tissue | From randomization (month 0) to 12 months
  Measurement of enzymes involved in lipid storage. FACS to examine the cellular composition of the adipose tissue sample and to allow downstream PCR analysis of DNA/RNA or western blot analysis of proteins from specific cell populations or from non-sorted biopsy material.
Explorative analysis of skeletal muscle tissue | From randomization (month 0) to 12 months
  FACS to examine the cellular composition and to allow downstream PCR analysis of DNA/RNA or western blot analysis of proteins from specific cell populations or from non-sorted biopsy material. RNA sequencing, and protein content will be assessed as metabolomics and proteomics by mass-spectrometry.
Whole body metabolism | From randomization (month 0) to 12 months
  Changes in circulating metabolic markers
Muscle metabolism | From randomization (month 0) to 12 months
  Changes in metabolic signature of muscle tissue assessed by liquid chromatography-high-resolution mass spectrometry
Skeletal muscle satellite cell (MuSC) proliferation assays | From randomization (month 0) to 12 months
  Proliferation and differentiation analysis in cell numbers and cell viability of MuSC

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wiggers, DMSC PHD MD, Principal Investigator — Dept. of Cardiology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thorup CV, Jeppesen CNA, Jensen TH, Tinggaard AB, Hvas CL, Rud CL, Skou MK, Mortensen JK, Reggiori F, Dengjel J, Wang J, Farup J, Jessen N, Kim WY, Wiggers H. POLYamine treatment in elderly patients with Coronary Artery Disease (POLYCAD): study protocol for a Danish randomised, double-blind, placebo-controlled trial of spermidine treatment versus placebo. Trials. 2025 Oct 30;26(1):452. doi: 10.1186/s13063-025-09176-z. PMID 41168834